CLINICAL TRIAL: NCT02944019
Title: Non-Interventional Study on Edoxaban Treatment in Routine Clinical Practice for Patients With Non Valvular Atrial Fibrillation
Brief Title: Edoxaban Treatment in Routine Clinical Practice for Patients With Non Valvular Atrial Fibrillation
Acronym: ETNA-AF-EU
Status: Completed | Type: Observational
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: DSE-EDO-04-14-EU
Record Dates: First submitted 2016-10-24; First posted 2016-10-25 (Estimated); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Atrial Fibrillation
Keywords: Nonvalvular Atrial Fibrillation; Post Authorisation Safety Study; Safety; Real World Evidence
MeSH Terms: conditions — Atrial Fibrillation | interventions — edoxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Edoxaban: Patients with established Non Valvular Atrial Fibrillation (NVAF) treated with edoxaban according to Summary of Product Characteristics (SmPC). Physician's prescribing behaviour will not be influenced, patients may only be included after the treating physician has made the clinical decision to prescribe edoxaban.
  Interventions: Drug: Edoxaban

INTERVENTIONS:
Drug: Edoxaban — Prescribed according to approved label
  Other Names: Lixiana

SUMMARY:
In order to understand the risks and benefits of edoxaban use in a real-world clinical setting in the Non-valvular Atrial Fibrillation (NVAF) indication, Daiichi-Sankyo proposed this post-authorization safety study (PASS) to gain insight into the safety (bleeding, liver adverse events, all-cause mortality and other drug related adverse events) of edoxaban use in patients with NVAF who were not preselected.

DETAILED DESCRIPTION:
Patients will be from 10 different European countries and care settings (primary and secondary care and different specialties). A one-year patient recruitment period per country is planned, but it could be longer if patient recruitment numbers are not reached. Patient data will be documented at baseline (BL), one annual data documentation point during the four-year follow up (FU), and at final assessment. Patients who permanently discontinue edoxaban during the observation period will continue to be followed annually for a further two years, or until the end of the observational period (whichever comes first).

ELIGIBILITY:
Inclusion Criteria:

* NVAF-patients treated with edoxaban according to Summary of Product Characteristics (SmPC).
* Written informed consent for participation in the study (ICF).
* Not simultaneously participating in any interventional study.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with NVAF and treated with edoxaban according to Summary of Product Characteristics (SmPC).
Sampling Method: Non-Probability Sample
Enrollment: 13980 (Actual)
Dates: Start 2015-08; Primary Completion 2022-04-13 (Actual); Study Completion 2022-04-13 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Experiencing Real-World Safety Data Events within 4 Years | within 4 years
  Real-world safety data events include bleeding events including intracranial haemorrhage, drug related adverse events such as liver adverse events, cardiovascular (CV) and all-cause mortality

SECONDARY OUTCOMES:
Percentage of Participants with Patient Relevant Outcomes | within 4 years
  Patient relevant outcomes include Strokes (ischaemic and haemorrhagic) , Systemic Embolic Events (SEE), Transient Ischemic Attack (TIA), Major Adverse Cardiovascular Events (MACE), Venous Thromboembolism (VTE), Acute Coronary Syndrome (ACS), and Hospitalisations related to a CV condition.
Percentage of Participants Compliant with Edoxaban Therapy | over 4 years
  Categories: Always, Almost Always, Most of the Time, Less than Half the Time, Unknown

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (724):
- Austria (23):
  - Wahlarzt Ordination, Dr. Paul Pinter, Altenmarkt, Altenmarkt
  - Krankenhaus St. Josef Braunau, Innere Medizin 2, Braunau, Braunau am Inn
  - Landeskrankenhaus Feldkirch, Kardiologie, Feldkirch, Feldkirch
  - Universitaetsklinik Graz, Onkologie, Graz, Graz
  - KRAGES Burgenlaendische Krankenanstalten LH Guessing, Innere Medizin, Guessing, Güssing
  - Klinikum Klagenfurt, Kardiologie, Klagenfurt, Klagenfurt
  - A. Oe. Kh Der Barmherzigen Schwestern, Kardiologie, Linz, Linz
  - Kepler Universitaetsklinikum, Kardiologie, Linz, Linz
  - Krankenhaus der Elisabethinen Linz, Kardiologie, Linz, Linz
  - Kepler Universitätsklinikum, Neurologie, Linz, Linz
  - Krankenhaus der Barmherzigen Brueder, Innere Medizin, Linz, Linz
  - Reha Zentrum Muenster, Neurologie, Muenster, Müenster
  - Dr. Peter Kaserer, Salzburg, Salzburg
  - Ordination Dr Kober, Sankt Aegyd am Neuwalde, Sankt Aegyd am Neuwalde
  - LKH Steyr, Kardiologie, Steyr, Steyr
  - AKH - Medizinische Universitaet Wien, Pulmomologie, Wien, Vienna
  - Allgemeines Krankenhaus Medizinische Universitaet Wien, Kardiologie, Wien, Vienna
  - Allgemeines Krankenhaus Medizinische Universitaet Wien, Unfallambulanz, Wien, Vienna
  - Universitaetsklinikum Wien, Neurologie, Wien, Vienna
  - Gruppenpraxis Dr. Scok, Wien, Vienna
  - Wilhelminenspital der Stadt Wien,Kardiologie,Wien, Vienna
  - Internistisches Zentrum Brigittenau, Innere Medizin, Wien, Vienna
  - LKH Villach, Innere Medizin, Villach, Villach
- Belgium (50):
  - Algemeen Stedelijk Ziekenhuis Campus Aalst, Cardiology, Aalst, Aalst
  - O.L.V Ziekenhuis, Aalst
  - Cliniques du Sud-Luxembourg, Cardiology, Arlon, Arlon
  - Huisartsenpraktijk Vileyn Bvba,Blankenberge, Blankenberge
  - Imeldaziekenhuis, Cardiology, Bonheiden, Bonheiden
  - A.Z. KLINA, Cardiology, Brasschaat, Brasschaat
  - AZ Sint-Jan Brugge, Cardiology 1, Brugge, Bruges
  - AZ Sint-Lucas, Cardiology, Brugge, Bruges
  - Clinique St-Jean, Cardiology, Bruxelles, Brussels
  - CHU Brugmann, Cardiology, Bruxelles, Brussels
  - CHU Brugmann, Neurology, Bruxelles, Brussels
  - Cliniques de l'Europe-St-Michel, Cardiology, Brussels, Brussels
  - Hopital Erasme, Cardiology, Bruxelles, Brussels
  - Universitair Ziekenhuis Brussel, Cardiology, Bruxelles, Brussels
  - Europa Ziekenhuizen, Cardiology, Brussel, Brussels
  - Private Practice Cardiology Dr Hollanders, De Pinte, De Pinte
  - AZ Sint-Blasius, Cardiology, Dendermonde, Dendermonde
  - UZ Antwerpen, Cardiology 1, Edegem, Edegem
  - UZ Antwerpen, Cardiology 2, Edegem, Edegem
  - A. Z. St-Dimpna, Cardiology, Geel, Geel
  - Ziekenhuis Oost Limburg, Cardiology, Genk, Genk
  - AZ Sint-Lucas - Campus Sint-Lucas, Gent, Ghent
  - Universitair Ziekenhuis Gent, Cardiology 1, Gent, Ghent
  - Universitair Ziekenhuis Gent, Neurology 1, Gent, Ghent
  - GHDC-Site Saint-Joseph, Cardiology, Gilly, Gilly
  - Private Practice Dr. Calozet, Gribomont, Gribomont
  - Jessa Ziekenhuis - Campus Virga Jesse, Cardiology, Hasselt, Hasselt
  - Jessa Ziekenhuis, Cardiology, Hasselt, Hasselt
  - St-Franciskus Ziekenhuis, Cardiology, Heusden-Zolder, Heusden-Zolder
  - Centre Hospitalier Hutois, Cardiology, Huy, Huy
  - AZ Zeno, Cardiology, Knokke-Heist, Knokke-Heist
  - AZ Groeninge - Campus Kennedylaan, Cardiology, Kortrijk, Kortrijk
  - AZ Groeninge Campus Loofstraat, Cardiology, Kortrijk, Kortrijk
  - VZW Regionaal Ziekenhuis Jan Yperman, Cardiology, Leper, Leper
  - UZ Leuven, Cardiology, Leuven, Leuven
  - CHR de la Citadelle, Cardiology, Liège, Liège
  - CHC-Clinique St-Joseph, Cardiology, Liège, Liège
  - AZ Sint-Maarten, Cardiology, Mechelen, Mechelen
  - CHU de Charleroi, Cardiology,Charleroi, Montigny-le-Tilleul
  - Centre de Cardiologie du Bauloy, Chevalier, Ottignies, Ottignies-Louvain-la-Neuve
  - Maria Ziekenhuis Noord-Limburg VZW, Cardiology, Overpelt, Overpelt
  - AZ Delta, Cardiology, Roeselare, Roeselare
  - AZ Glorieux, Cardiology, Ronse, Ronse
  - AZ Nikolaas, Cardiology, Sint-Niklaas, Sint-Niklaas
  - AZ Turnhout - Campus Sint-Elisabeth, Cardiology, Turnhout, Turnhout
  - Private Practice Cardiology Dr Huisartsen Dierickx, Westouter, Westouter
  - BVBA Cardiology Dr. Luc Capiau, Wetteren, Wetteren
  - Practice Dr. Axel Caenepeel, Willebroek, Willebroek
  - CHU UCL Namur - Mont-Godinne, Cardiology, Yvoir, Yvoir
  - St Elisabeth Ziekenhuis, Cardiology, Zottegem, Zottegem
- Germany (304):
  - Praxis für Kardiologie Aachen GbR, Aachen
  - Praxis Dr. Stephan Keldenich, Aachen
  - Innere Medizin im Gesundheitszentrum, Ahrensburg
  - Gemeinschaftspraxis Dres. Franz Gaim & Peter Anton, Aiterhofen
  - Prof. Dr. Med. Karl Josef Osterziel und Peter Wittmann Oberpfalz GbR, Amberg
  - Gemeinschaftspraxis Dr. Med. Sylvia Baumbach und Dr. Elke Reichelt, Apolda
  - Ilm-Kreis-Kliniken Arnstadt-Ilmenau gGmbH, Arnstadt
  - Praxis Dr. Wende, Aschaffenburg
  - Praxis N. Nabo/H.J. Dworatzek, Bad Abbach
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Herz-Kreislauf-Klinik Bevensen AG, Bad Bevensen
  - Praxis Dr. Med. Wildenauer, Bad Brückenau
  - Praxis Prof. Dr. Med. Emanuel Fritschka, Bad Brückenau
  - Praxis Dr. Med. Vivion Koppatsch, Bad Buchau
  - SLK-Kliniken Heilbronn GmbH Klinikum am Plattenwald, Bad Friedrichshall
  - Herzcarre Kardiologie Bad Homburg, Bad Homburg
  - Kardiologische Praxis Dr. Med. Wolfgang Jungmair, Bad Homburg
  - Praxis Dr. Med. Detlef Hammerschmidt, Bad Krozingen
  - Praxis Dres. Fissan und Werner, Bad Lippspringe
  - Kerckhoff-Klinik GmbH - Abt. Administration Forschung und Lehre, Bad Nauheim
  - Sportklinik Bad Nauheim, Bad Nauheim
  - Rhön-Klinikum AG, Rhön-Klinikum Campus Bad Neustadt, Bad Neustadt an der Saale
  - Praxis Dr. Med. Zimny, Bad Pyrmont
  - Praxis Dr. Jenniches, Bad Salzdetfurth
  - Praxis am Landratspark, Bad Segeberg
  - Praxis Dr. Med. Venesa Hild, Bad Soden-Salmünster
  - Praxis Dr. Med. Karl-Heinz Schnaibel, Baden-Baden
  - Kariologische Gemeinschaftspraxis Mosbach Dres. Haney/Gehrig/Loges, Baden-Württemberg
  - Praxis Georg Behnes, Baden-Württemberg
  - Gemeinschaftspraxis Dr. Patrick Abdul-Malak & Reinhard Lieb, Bahrdorf
  - Gemeinschaftspraxis Dres. Seitz und von Meißner, Baiersbronn
  - Praxis Dr. Med. Ulrich Jäck, Balingen
  - Cims Ug Mbh, Bamberg
  - Gemeinschaftspraxis PD Dr. Med. Bernd Hammer und Alexander Schilling, Bechhofen
  - Hausärztliche-Internistische Praxis Dr. Med. Gerd-Ulrich Heinz, Bergisch Gladbach
  - KardioPraxis - Gemeinschaftspraxis für Herz-Kreislauferkrankungen, Bergisch Gladbach
  - Kardiologische Praxis Dr. Med. Sabine Roeder, Berlin
  - Praxisgemeinschaft Rankestrasse, Berlin
  - Charité - Universitaetsklinikum Berlin - Campus Benjamin Franklin, Berlin
  - MVZ Gropiusstadt, Berlin
  - Praxis Dr. Med. Andreas Kopf, Berlin
  - Kardiologische Facharztpraxis Dr. Anne Winkelmann, Berlin
  - Herzpraxis Hohenschönhausen, Berlin
  - DRK Kliniken Berlin Westend, Berlin
  - Gemeinschaftspraxis Dres. Frank Eickhoff und Jan Lokies, Berlin
  - Internistische Gemeinschaftspraxis Biedenkopf, Biedenkopf
  - Marienhaus Klinikum Eifel Bitburg, Bitburg
  - Praxis Dr. Med. Annette Biedermann, Blankenhain
  - Praxis Dr. Med. Sabine Lorenz, Bochum
  - Praxis Dr. med. Ulrike Spengler, Borsdorf
  - Städtisches Klinikum Brandenburg, Brandenburg
  - Kardiologie an der Paulikirche, Braunschweig
  - Fürst-Stirum-Klinik Bruchsal, Bruchsal
  - Kardiologie im Friedrichspalais, Bruchsal
  - Praxis Dr. Med. Fabian Schmidtler, Burghausen
  - Medizinisches Versorgungszentrum am Küchwald GmbH, Chemnitz
  - Kardiologische Gemeinschaftspraxis Dres. Kaltofen / Schubert / Gerner/ Jurowsky, Chemnitz
  - Kardiologische Praxis Dr. Med. Steffen Tröger, Chemnitz
  - Praxis für Innere Medizin und Kardiologie - Dipl.-Med. Karl-Heinz Schermaul, Chemnitz
  - Kardiologische Praxis Dr. Med. Heiko Stellmach, Chemnitz
  - St. Josefs-Hospital, Cloppenburg
  - Klinikum Coburg GmbH, Coburg
  - Kardiologie Fritsch - Facharztzentrum am Heilig Geist-Gesundheitszentrum, Cologne
  - Praxis für Innere Medizin, Kardiologie, Pneumologie, Cologne
  - MVZ im Rolshover Hof AmKaRe Poll - Dres. Gysan, Heinzler, May GbR, Cologne
  - HELIOS Amper-Klinikum Dachau, Dachau
  - Praxis Dr. Rolf Dietzel und Kollegen - ortsübergreifende Gemeinschaftspraxis, Dannenfels
  - Praxis Raphael Steger, Deggenhausen
  - Praxis für Allgemeinmedizin Dr. Med. Günter Häfele, Denzlingen
  - Praxis für Kardiologie und Angiologie Dr. Med. Frank Menzel, Dessau
  - Gemeinschaftspraxis Dr. Med. Reinhold Jerwan-Keim, Renate Metz, Dietzenbach
  - Praxis für Kardiologie, Gesundheitsförderung und Prävention, Dormagen
  - Praxis Dr. med. Jan-Gerrit Voigt, Dorsten
  - Kardiologische PraxisGemeinschaft Kampstraße, Dortmund
  - Klinikum Dortmund gGmbH, Dortmund
  - Gemeinschaftspraxis für Kardiologie Dr. med. Thomas Wetzel und Dr. Sebastian Willgeroth, Dortmund
  - Allgemeinarztpraxis im PueD, Dortmund
  - Praxis Dr. Med. Binder, Dreieich
  - Zentrum für klinische Prüfungen in der Facharztzentrum Dresden-Neustadt GbR, Dresden
  - Praxisklinik Herzkreislauf am Wasa-Platz, Dresden
  - Hausärztlich-Kardiologisches MVZ, Am Felsenkeller" GmbH, Dresden
  - Kardiologen am Fetscherplatz - Gemeinschaftspraxis für Kardiologie Dr. Med. Michael Günther & Dr. Med. Steffen Kolschmann, Dresden
  - Technische Universität Dresden, Dresden
  - Universitätsklinikum Carl Gustav Carus TU Dresden, Dresden
  - Gemeinschaftspraxis Alain Barakat und Helene Willems, Duisburg
  - Evangelisches Krankenhaus Düsseldorf, Düsseldorf
  - Praxis Dres. Rolfes & Schapfeld, Egelsbach
  - Praxis Dipl.- Med. Petra Herrmann, Eisenach
  - Berufsausübungsgemeinschaft Holger Michel und Franziska Leffler, Eisleben Lutherstadt
  - Praxis Dr. Med. Andreas Hagenow, Elsterwerda
  - Kreiskrankenhaus Emmendingen, Emmendingen
  - Internistische Schwerpunkt Praxen, Erlangen
  - Überörtliche Gemeinschaftspraxis Dres. Kessler, Kessler-Schwigon & Kollegen, Erlangen
  - Praxis Dr. Schmitz, Erlenbach
  - Gemeinschaftspraxis Hanfstingl, Erlensee
  - Gemeinschaftspraxis Dres. Hagemann, Dürfeld und Breiderhoff, Essen
  - Praxis am Markt, Essen
  - Studienzentrum Bocholderstrasse, Dres. Med. Faghih/Zühlke, Essen
  - Praxis Dr. Med. Thomas Ludwig, Farchant
  - DIAKO Krankenhaus gGmbH, Flensburg
  - Praxis für Herz-Kreislauf Erkrankungen, Flensburg
  - Praxis Dres. Fabian Tölle und Bernadette Jauch GbR, Flieden
  - Internistische Gemeinschaftspraxis Dr. Med. Engelhard / Dr. Med. Wihl, Frankenberg
  - Kardiocentrum Frankfurt an der Klinik Rotes Kreuz, Frankfurt
  - Dipl.- Med. Kerstin Steinbach, Freital
  - Bürgerhospital Friedberg Neurologie, Friedberg
  - Gemeinschaftspraxis Dres. Simon, Schwuchow, A. u. C. Hölscher, I. Olbert und M. Conze, Fulda
  - Gemeinschaftspraxis im Altstadt-Carree Dres. Simon, Schwuchow, A. u. C. Hölscher, I. Olbert und M. Conze, Fulda
  - Kardiologische Gemeinschaftspraxis Gelsenkirchen, Gelsenkirchen
  - Gemeinschaftspraxis Dr. Med. Hans-Walter Bindig und Carl-André Bystron, Georgensgmünd
  - Praxis Dr. Med. Christian Oehlwein, Gera
  - Praxis für Kardiologie Dr. Med. Jörg Langel, Gera
  - Gemeinschaftspraxis Dr. Unger und Zawalski, Giengen an der Brenz
  - Kardiologische Praxis Dr. Med. Frank Warzok, Gotha
  - Praxis Dr. Med. Karsten Müller, Gräfenhainichen
  - Gemeinschaftspraxis Dres. Hetzel & Grewe-Kemper, Greven
  - DRK-Krankenhaus Grevesmühlen gGmbH, Grevesmühlen
  - Kardiologische Praxis Dr. Tauchert und Prof. Dr. Warnholtz, Griesheim
  - Praxis Carlo Buttron, Groß-Rohrheim
  - Praxis Dr. Med. Peter W. Frank, Gröbenzell
  - Klinikum Gütersloh gGmbH, Gütersloh
  - Hausarztpraxis und Diabetologische Schwerpunktpraxis Dr. Med. Jörg A. Hintze und Dr. Med. Martin Grundner, Hainburg
  - Praxis Dr. Dubiel, Hamburg
  - Medizinisches Versorgungszentrum für Innere Medizin, Hamburg
  - Praxis Dr. Brauer, Hamburg
  - Praxisgemeinschaft Oldesloer Strasse, Dr. med. Johannes Spormann, Hamburg
  - Kardiologie am Tibarg, Hamburg
  - Ärztezentrum Hammelburg / Dres Edgue/Barbuia/Linke, Hammelburg
  - Gemeinschaftspraxis Ewa Drzewinska und Dr. Magdalena ten Hoevel, Hamminkeln
  - Praxis Andre Terhorst, Hamminkeln
  - Praxis Dr. Med. Glatzel, Hanover
  - Hassberg-Kliniken Haus Hassfurt, Haßfurt
  - Kardiologische Praxis Holger Killat, Haßloch
  - Atos Klinik Heidelberg, Heidelberg
  - Heidelberger Praxisklinik für Innere Medizin, Kardiologie und Pneumologie, Heidelberg
  - Kardiologische Schwerpunktpraxis, Heidelberg
  - Praxis für Angiologie und Hämatologie Dr. Med. Bernadett Brado, Heidelberg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Praxis Dr. Med. Rainer Droste, Heilbronn
  - Praxis Dr. Med. Nils Jonas, Heitersheim
  - Kardiologie Alsterquelle, Praxis Dr. Jörg Kynast, Henstedt-Ulzburg
  - Klinikum Herford, Herford
  - Praxis Dr. Wolfgang Albrecht, Heusenstamm
  - Kardiologische Praxis Winkler, Hohenstein-Ernstthal
  - Universitätsklinikum des Saarlandes, Homburg
  - Praxis Dr. Med. Josef Lißmann, Homburg
  - Praxis Dr. Med. Susanne Schöller, Horb
  - iKardio, Hürth
  - Gemeinschaftspraxis Dr. Med. Paul Hegemann / Dr. Med. Claus Franck, Ingelheim
  - Kardio-IN - Kardiologische Gemeinschaftspraxis Ingolstadt, Ingolstadt
  - Universitätsklinikum Jena, Jena
  - Praxisgemeinschaft Jerichow, Jerichow
  - St. Elisabeth Krankenhaus Jülich, Jülich
  - Westpfalz-Klinikum GmbH - Standort I, Kaiserslautern
  - Praxis Dr. Med. Hermann Burkei, Kaiserslautern
  - Praxis Dr. Med. Joachim Heisters, Kamp-Lintfort
  - Internistisch-Kardiologische Praxis Kandel, Kandel
  - SRH Klinikum Karlsbad-Langensteinbach GmbH, Karlsbad
  - Kardiologische Praxis Waldstraße, Karlsruhe
  - Kardiologie Gemeinschaftspraxis Kassel, Kassel
  - B. Braun Cardio Zentrum Kassel MVZ GmbH, Kassel
  - Berufsausübungsgemeinschaft Dres. Med. Kolitsch / Müller, Katzhütte
  - Klinikum Konstanz, Konstanz
  - Gemeinschaftspraxis Dres. Persicke und Scheuermann, Kornwestheim
  - Praxis Dr. Matthias Claus, Köpenick
  - Kardiologische Praxis Dres. Rieber and Ganschow, Leinfelden-Echterdingen
  - Kardiologische Gemeinschaftspraxis Dres. Loebe, Weißbrodt, Leipzig
  - Universitätsklinikum Leipzig AöR, Leipzig
  - Klinikum St. Georg gGmbH, Leipzig
  - Herzzentrum Leipzig GmbH, Leipzig
  - Praxis am Oberen Tor Dr. med. Ilka Simon-Wagner, Lichtenfels
  - Praxisgemeinschaft Dr. H. Boeneke / R. P. Vormann, Lienen
  - Gemeinschaftspraxis Dres. Med. Pfeffer · Sauer · Eiser, Lindenberg
  - Praxisgemeinschaft Dr. Biesenbaum und Dr. Gerbaulet, Löhne
  - Cardio Centrum Ludwigsburg Bietigheim, Ludwigsburg
  - Praxis Dr. Med. Achim Ulmer, Ludwigsburg
  - Praxis Dr. Med. Hannelore Pitule, Ludwigshafen
  - Kardiologische Praxisklinik Ludwigshafen, Ludwigshafen
  - Praxis Dr. Med. Jörn Weckmüller, Lübeck
  - SANA Klinik Lübeck, Lübeck
  - Gemeinschaftspraxis Erdmann Schütz, Lünen
  - Universitätsklinikum Magdeburg A.ö.R., Magdeburg
  - Cardiopraxis Mainz und Ingelheim GbR - MED Facharztzentrum, Mainz
  - Katholisches Klinikum Mainz, Caritas Werk St. Martin Gem. Träger und Betriebsf. GmbH, Mainz
  - Gemeinschaftspraxis Vogelstang, Mannheim
  - Kardiologische Praxis Dr. Jens Taggeselle, Markkleeberg
  - Praxis Dr. Med. Stephan Kreutz, Maxdorf
  - Praxis für Allgemeinmedizin, Großes Palais Meiningen - Das Ärzte- und Gesundheitszentrum, Meiningen
  - Internistisches Facharztzentrum mit Dialyse Fachbereich Kardiologie - Angiologie, Memmingen
  - Carl-von-Basedow-Klinik Saalekreis GmbH, Merseburg
  - Praxis Dr. Matthias Läger, Merseburg
  - Überörtliche Berufsausübungsgemeinschaft - Dres. Med. Beate Zygan, Thomas Reiff, Stephan Linse, Afif Haj-Yehia, Moers
  - Herz-/ Gefäßpraxis Morsbach am Teufelsbrunnen, Morsbach
  - Institut für Hämostaseologie GmbH, Möser
  - Praxis Dr. Med. Andreas Gammel, Mössingen
  - Praxis Dr. Kai-Alexander Dähmlow, Murrhardt
  - Gemeinschaftpraxis Dr. Med. Martin Prohaska und Dr. Med. Felix Schulte, Mühldorf
  - Kardiologie Mühldorf am Inn Dr. Med. Norbert Schön, Mühldorf
  - Kardiologie am Rotkreuzplatz, München
  - Kardiologische Gemeinschaftspraxis an der Universität Dr. Med. Wauer und Dr. Med. Windstetter, München
  - Klinikum der Universität München, München
  - München Klinik gGmbH - Klinikum Neuperlach, München
  - Praxis für Innere Medizin, Münster
  - Gefäßzentrum Dr. Heckmann und Kollegen, Neckargemünd
  - Praxis Dr. Alex Berinde, Neu-Isenburg
  - Dr. Klimek MVZ GmbH, Neuburg an der Donau
  - Hausärztliche Praxisgemeinschaft Dr. Med. Roland Krämer und Dr. Med. Peter Rauh, Neukölln
  - Praxis Dr. Falkenstein and Dr. Löser, Neustadt
  - Marienhaus Klinikum Neuwied, Neuwied
  - Gemeinschaftspraxis Dres. Med. Hartwig & Henrik Schumann, Nidderau
  - Kardiologische Praxis Nienburg, Nienburg
  - Gemeinschaftspraxis Prof. Dr. Med. N. Ludwig & Dr. Med. B. Honl, Nordheim
  - Kardiologische Praxis Northeim, Northeim
  - Kardiologie am Weißen Turm Dr. Med. Alexander Stadelmann, Nuremberg
  - Innere am Stadtpark, Nuremberg
  - Praxis Dr. Med. Yuriy Amdur, Nuremberg
  - Gemeinschaftspraxis Dres. Med. Barth, Birkofer, Müller-Hörner, Schwab, Nuremberg
  - Medic Center Nürnberg, Nuremberg
  - MCN Medic-Center Nürnberg GmbH, Nuremberg
  - Praxen Dr. Bögel, Völk und Kollegen, Nuremberg
  - Martha Maria MVZ, Praxis Kardiologie, Nuremberg
  - Krankenhaus Martha-Maria Nürnberg, Nuremberg
  - Praxis Dr. Med Udo Frädrich, Oberhausen
  - Praxis Dr. Med. Gunter Hergdt, Obermichelbach
  - Praxis Dr. Med. Bachhuber, Oberndorf
  - Gemeinschaftspraxis Klaus Peter Dausend und Joachim Hock, Obernkirchen
  - Hausarztpraxis-Offenbach, Offenbach
  - Praxis Dr. Med. Lutz Kröning, Offenbach
  - Praxis Drs Wiese/Metreveli-Wiese, Osnabrück
  - St. Vincenz-Krankenhaus GmbH, Paderborn
  - Kardiologische Praxis Papenburg Dr. Andreas Wilke & Dr. Andrej Malazhavy, Papenburg
  - MVZ Birkenallee GmbH, Papenburg
  - MVZ DaVita Kardiologisches Zentrum Peine GmbH, Peine
  - Praxis Dr. Med. Karl Bruck, Pirmasens
  - Hausärztlich-Kardiologisches MVZ "Am Felsenkeller" GmbH, Pirna
  - Kardiologische Gemeinschaftspraxis am Park Sanssouci, Potsdam
  - Praxis S. Tlechas-Tkatsch, Potsdam
  - Harzklinikum Dorothea Christiane Erxleben GmbH, Quedlinburg
  - Paracelsus-Harz-Klinik Bad Suderode GmbH, Quedlinburg
  - Allgemeinmedizinisch Internistische Praxis Dr. Med. Harald Borgmann, Radebeul
  - Gemeinschaftspraxis Dr. med. Bruno Kronschnabl, Dr. Med. Manuel Kronschnabl, Sonja Römer-Kronschnabl, Regen
  - Kardiologische Gemeinschaftspraxis Dr. med. Kösler, Dr. Med. Bauer, Dr. Med. Buresch und Prof. Dr. Med. Niederer, Regensburg
  - Gemeinschaftspraxis Dres. Klein, Schreiber, Remagen
  - Kardiologische Gemeinschaftspraxis RT, Reutlingen
  - Herz Riesa - Gemeinschaftspraxis Dres. Med. Stenzel, Ebert & Otto, Riesa
  - Praxis Dr. Med. Stefan Schneider, Rieschweiler-Mühlbach
  - Praxis für Allgemeinmedizin Dr. Loeseken, Rohrberg
  - Universitätsmedizin Rostock, Rostock
  - Herz- und Kreislauf-Zentrum Rotenburg a. d. Fulda, Rotenburg an der Fulda
  - Dres. Med. Claudia Wankmüller u. Michael Dusold, Rottweil
  - Praxis Dr. Med. Andreas Ecke, Rottweil
  - Praxis Dr. Med. Thomas Pätzold, Rudolstadt
  - MVZ MP Saaletal, Saalfeld
  - Praxisklinik Salzatal, Salzmünde
  - Gemeinschaftspraxis Dres. Michael Eis und Günter Rehling, Sand
  - Gemeinschaftspraxis Amin Satli und Dr. Med. Bernd Schüttrumpf, Sarstedt
  - Praxisgemeinschaft Jerichow, Schönhausen
  - Praxis Dr. Robert Tecl & Kollegen, Schriesheim
  - Asklepios Klinikum Schwalmstadt, Schwalmstadt
  - Praxis Dr. H.-J. Scholz, Schwetzingen
  - Zentrum für Prävention und Rehabilitation, Praxisgemeinschaft Dr. Med. Ulrich Overhoff, Dr. Med. Fabian Krämer, Siegen
  - Diabetologische Schwerpunktpraxis Dres. Segiet, Gleixner und Bode, Speyer
  - Diakonissen-Stiftungs-Krankenhaus Speyer, Speyer
  - Praxis Prof. Staedt / Dr. Med. M. Münchbach, Speyer
  - Parkkardiologie, Stahnsdorf
  - Hausarztpraxis W. Wagner und Dr. E. Hofmann, Stegaurach
  - Johanniter-Krankenhaus Genthin - Stendal gGmbH, Stendal
  - Praxis Dr. Med. Annette Birkenhagen, Stolberg
  - Internistische Gemeinschaftspraxis Steiner Thor, Straubing
  - Praxis Dres. Wolf, Straubing
  - Überörtliche Berufsausübungsgemeinschaft Dres. Med. Knöbel / Pelz-Knöbel / Olesch / von Hassel / Spaltmann, Straubing
  - Ärztehaus Kastanienallee - Praxis Dr. Michael Rother, Strausberg
  - Klinikum Stuttgart, Stuttgart
  - Kardiologische Gemeinschaftspraxis Dres Klein & Neumann, Stuttgart
  - Praxis Dr. Mirko Böhme, Sulzberg
  - Kreiskrankenhaus Torgau "Johann Kentmann" gGmbH, Torgau
  - Praxis Dr. Med. Astrid Schmidt-Reinwald, Trier
  - Agaplesion Bethesda Klinik Ulm, Ulm
  - Herzklinik Ulm, Dr. Haerer und Partner, Ulm
  - Universitätsklinikum Ulm, Ulm
  - Praxis Dr. Med. Roland Braun, Unterschneidheim
  - Praxis Dr. Med. Sabine Hansen, Unterwellenborn
  - Hausarzt-Praxis Dr. Thomas Hohenstatt Dr. Med. Antonia Dengler, Ursensollen
  - Praxis im Alten Rathaus, Einzelpraxis Dr. Med. R. Berg, Ühlingen-Birkendorf
  - Schwarzwald-Baar Klinikum Villingen-Schwenningen GmbH, Villingen-Schwenningen
  - INNERE MED3 - Praxis für Innere Medizin, Walldorf
  - Praxis Georg Weiß, Weingarten
  - Kardiologische BAG - Dr. med. Glatthor, Dr. Med. Müller, Dr. Med. Schlotterbeck und Dr. Med. Trompler, Weingarten
  - Praxis Sigmund Jakob, Weinsberg
  - Internistische Praxis Hugo Loeber, Weiskirchen
  - Internistische Gemeinschaftspraxis Thomas A. Sanner & Uwe Wojts, Weißenstadt
  - Kardiologische Praxis Dr. Al-Zoebi, Wermsdorf
  - Praxis Karsten Becker, Wesel
  - Praxis H. Aslan, Wetzlar
  - Hausarztpraxis Anna Lorenz und Detlef Germann, Wetzlar
  - Praxis Dr. Med. Reinhold Schneider und Christine Schneider, Wetzlar
  - Internistische Praxisgemeinschaft, Weyhe
  - Praxis für Innere Medizin Tunca Karakas, Wiesbaden
  - Praxis Abdel-Qader, Winsen
  - Praxis Dr. Med. Eißfeller, Wöllstein
  - Praxis Dr. Tripathi, Wuppertal
  - Universitätsklinikum Würzburg, Würzburg
  - Praxis Jürgen Krafft, Zirndorf
  - INFO-MED Leipzig GmbH, Zwenkau
- Ireland (10):
  - Cork University Hospital, Cardiology, Cork, Cork
  - Mater Misericordiae University Hospital, Respiratory Medicine, Dublin, Dublin
  - St. James's Hospital, Dept. of Cardiology, Dr. Ross T. Murphy, Dublin, Dublin
  - Beacon Hospital, Cardiology, Dublin, Dublin
  - Beaumont Hospital, Cardiology, Dublin, Dublin
  - University Hospital Galway, Cardiology, Galway, Galway
  - St. Luke's General Hospital, Cardiology, Kilkenny, Kilkenny
  - Letterkenny General Hospital, Cardiology, Letterkenny, Letterkenny
  - University Hospital Limerick, Cardiology, Co Limerick, Limerick
  - Our Lady's Hospital, Dept. of Medicine, Dr Mazen Al Alawi, Navan, Navan
- Italy (170):
  - Casa di cura privata Villa dei Fiori srl, Acerra
  - Ospedale Generale Regionale "F. Miulli", Acquaviva delle Fonti
  - ASL AL Presidio Ospedaliero SS Antonio e Biagio e Cesare Arrigo, Alessandria
  - A.O.U. Ospedali Riuniti Umberto I - G.M. Lancisi - G. Salesi, Ancona
  - Istituto Nazionale di Riposo e Cura per Anziani IRCCS, Ancona
  - Ospedale Civile Lorenzo Bonomo, Andria
  - Ospedale di Anzio- Nettuno-ASL Roma H, Anzio
  - Ospedale San Donato di Arezzo, Arezzo
  - Ospedale E.Muscatello - Augusta, Augusta
  - Azienda Ospedaliera di Rilievo Nazionale e di Alta Specialità San Giuseppe Moscati, Avellino
  - Ospedale San Paolo, Bari
  - Azienda Ospedaliero Universitaria Consorziale Policlinico, Bari
  - Casa di Cura Tricarico Rosano, Belvedere Marittimo
  - Azienda Ospedaliera Gaetano Rummo, Benevento
  - Ospedale Papa Giovanni XXIII - ASST Papa Giovanni XXIII, Bergamo
  - Ospedale Vittorio Emanuele II, Bisceglie
  - Ospedale Maggiore di Bologna AUSL di Bologna, Bologna
  - Azienda Ospedaliero Universitaria di Bologna Policlinico Sant'Orsola - Malpighi, Bologna
  - Ospedale di Bellaria AUSL di Bologna, Bologna
  - Ospedale di Bolzano, Bolzano
  - Ospedale "Santa Maria", Borgo Val di Taro
  - ASST Ospedale Spedali Civili, Brescia
  - Fondazione Poliambulanza Istituto Ospedaliero, Brescia
  - Ospedale S. Giovanni di Dio, Cagliari
  - Ospedale Brotzu di Cagliari, Cagliari
  - Ospedale "Gravina e Santo Pietro " Caltagirone, Caltagirone
  - Ospedale di Camposampiero - Ulss 6 Euganea, Camposampiero
  - Azienda Ospedaliera di Caserta, Sant'Anna e San Sebastiano, Caserta
  - Istituto Scientifico Ospedale Maugeri di Cassano delle Murge, Cassano delle Murge
  - Ospedale Santa Scolastica di Cassino-ASL di Frosinone, Cassino
  - Ospedale Unico della Valtidone, Castel San Giovanni
  - Presidio Ospedaliero Garibaldi-Nesima, Catania
  - Ospedale Ferrarotto Alessi di Catania, Catania
  - Ospedale Cannizzaro, Catania
  - A.O.U. Mater Domini, Catanzaro
  - Ospedale M. Bufalini, Cesena
  - ASL n. 2 Lanciano Vasto Chieti Ospedale SS. Annunziata di Chieti, Chieti
  - Ospedale di Chioggia - Ulss 3 Serenissima, Chioggia
  - Ospedale Bassini _ASST MI Nord, Cinisello Balsamo
  - Ospedale Civile di Ciriè, Cirié
  - Ospedale San Giuseppe Copertino, Copertino
  - Ospedale Santa Margherita - Valdichiana, Cortona
  - ASST Ospedale Maggiore di Crema, Crema
  - Ospedale di Cremona - ASST di Cremona, Cremona
  - Ospedale di Rete "Engles Profili", Fabriano
  - Arcispedale S. Anna, Ferrara
  - P.O. Vaio Fidenza - AUSL Parma, Fidenza
  - Ospedale Santa Maria Nuova di Firenze, Florence
  - A.O.U. Careggi, Florence
  - Azienda Ospedaliero Universitaria "Ospedali Riuniti" di Foggia, Foggia
  - Ospedale "Morgagni - Pierantoni" di Forlì, Forlì
  - Ospedale di Frascati, Frascati
  - Ospedale "Fabrizio Spaziani"-ASL di Frosinone, Frosinone
  - Ospedale Villa Scassi ASL GE 3 Genovese, Genova
  - IRCCS. A.O.U. San Martino IST, Genova
  - Ospedale Padre Antero Micone di Sestri Ponente - ASL 3 Genovese, Genova
  - Ospedale di Gorizia, Gorizia
  - P.O. di Grosseto, Grosseto
  - Ospedale Ferdinando Veneziale, Isernia
  - Presidio Ospedaliero di Latisana e Palmanova, Latisana
  - ASST Lecco - P.O. di Merate, Lecce
  - GVM - Città di Lecce Hospital, Lecce
  - Ospedale Vito Fazzi, Lecce
  - Poliambulatorio Cittadella della Salute, Lecce
  - ASST Ovest Milanese Ospedale Civile di Legnano, Legnano
  - Ospedali Riuniti di Livorno - USL Toscana nord ovest, Livorno
  - Ospedale San Salvatore, L’Aquila
  - Ospedale San Camillo De Lellis, Manfredonia
  - Ospedale di Mantova - ASST di Mantova, Mantova
  - Ospedale Paolo Borsellino di Marsala, Marsala
  - Ospedale Civile USL1 di Massa Carrara, Massa Carrara
  - ASM Matera Presidio Ospedaliero Madonna delle Grazie, Matera
  - Casa di Cura Privata Montevergine S.p.A., Mercogliano
  - A.O. Universitaria Policlinico " G. Martino" Messina, Messina
  - Ospedale dell'Angelo - ULSS 3 Serenissima, Mestre
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale San Raffaele, Milan
  - Centro Cardiologico Monzino, Milan
  - Istituto Scientifico Ospedale San Luca, Milan
  - Grande Ospedale Metropolitano di Niguarda, Milan
  - Presidio di Mirano - Ulss 3 Serenissima, Mirano
  - Policlinico di Modena, Modena
  - Nuovo Ospedale Civile S. Agostino-Estense, Modena
  - Regina Montis Regalis Mondovì_ASL CN 1, Mondovì
  - Ospedale San Giacomo di Monopoli, Monopoli
  - ASST Monza- Ospedale San Gerardo, Monza
  - Policlinico di Monza, Monza
  - Ospedale Riabilitativo di Motta di Livenza, Motta di Livenza
  - ASL NA 1 Presidio Ospedaliero Santa Maria di Loreto Mare, Napoli
  - Clinica Mediterranea SPA, Napoli
  - Ospedale Buon Consiglio Fatebenefratelli, Napoli
  - A.O.R.N. A. Cardarelli, Napoli
  - Azienda Ospedaliero Universitaria "Federico II", Napoli
  - Ospedale Monaldi - AOS dei Colli, Napoli
  - ASL NA 1 Centro P.O. dei Pellegrini, Napoli
  - Ospedale Classificato "Sacro Cuore - Don Calabria" di Negrar, Negrar
  - Ospedale Santa Maria della Pietà, Nola
  - Azienda Ospedaliero - Universitaria Maggiore della Carità, Novara
  - Ospedale S. Giacomo, Novi Ligure
  - Ospedale San Francesco di Nuoro, Nuoro
  - Policlinico San Marco, Osio Sotto
  - Azienda Ospedaliera di Padova, Padua
  - Buccheri La Ferla Fatebenefratelli, Palermo
  - Casa di Cura Candela, Palermo
  - A.O. Ospedali Riuniti Villa Sofia-Cervello, Palermo
  - Maria Eleonora Hospital di Palermo, Palermo
  - Ospedale della Media Valle del Tevere di Perugia, Pantalla
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Istituto di Cura Città di Pavia, Pavia
  - Centro Cuore Morgagni, Pedara
  - Azienda Ospedaliera di Perugia Ospedale S. Maria della Misericordia, Perugia
  - Ospedale Civile Spirito Santo, Pescara
  - Ospedale "Guglielmo da Saliceto", Piacenza
  - Ospedale S. Corona ASL 2 Savonese, Pietra Ligure
  - Ospedale Pieve di Coriano -ASST di Mantova, Pieve di Coriano
  - Ospedale Civile Edoardo Agnelli, Pinerolo
  - Azienda Ospedaliero Universitaria Pisana Cisanello, Pisa
  - Fondazione Toscana Gabriele Monasterio, Pisa
  - Nuovo Ospedale Santa Chiara, Pisa
  - AOR San Carlo, Potenza
  - Ospedale Santa Maria delle Grazie, Pozzuoli
  - Azienda USL Toscana Centro - Presidio "Misericordia e Dolce", Prato
  - Ospedale di Rho - ASST Rhodense, Rho
  - Ospedale "Infermi" di Rimini - AUSL Romagna, Rimini
  - Azienda Ospedaliera Ospedali Riuniti di Rivoli, Ospedale degli Infermi, Rivoli
  - Ospedale Policlinico Casilino, Roma
  - Ospedale G.B. Grassi-ASL Roma D, Roma
  - Policlinico dell'Università Campus Bio-Medico di Roma, Roma
  - Policlinico Tor Vergata, Roma
  - Ospedale San Filippo Neri-ASL Roma E, Roma
  - Ospedale S.Eugenio-ASL Roma C, Roma
  - Policlinico Umberto I, Roma
  - Istituto Dermopatico dell'Immacolata IDI-IRCCS, Roma
  - Fondazione Policlinico Universitaria "A.Gemelli", Roma
  - Ospedale San Giovanni Addolorata, Roma
  - Ospedale "San Giovanni Calibita" Fatebenefratelli Isola Tibertina, Roma
  - A.O. Sant'Andrea, Roma
  - Istituto Clinico Humanitas, Rozzano
  - Ospedale Orlandi di Bussolengo - ULSS 9 Scaligera, S. Bonifacio
  - A.O.U. OO.RR. San Giovanni di Dio Ruggi d'Aragona, Salerno
  - ULSS 9 Scaligera Presidio Ospedaliero Fracastoro, San Bonifacio
  - Ospedale di San Donà di Piave - ULSS 4 Veneto Orientale, San Donà di Piave
  - Ospedale S. Anna - ASST Lariana, San Fermo della Battaglia
  - Ospedale San Giovanni di Dio, San Michele
  - Ospedale Teresa Masselli Mascia, San Severo
  - Ospedale di Saronno - ASST Valle Olona, Saronno
  - ASL5 Liguria Ospedale San Bartolomeo, Sarzana
  - Ospedale SS. Annunziata di Sassari, Sassari
  - Ospedale Senigallia, Senigallia
  - ASST Bergamo EST Ospedale Bolognini, Seriate
  - Ospedale S.Rocco, Sessa Aurunca
  - Ospedale Le Scotte di Siena, Siena
  - ASST Valtellina e Alto Lario- Ospedale di Sondrio, Sondrio
  - Ospedale SS. Trinità-Sora, Sora
  - Ospedale Umberto I di Siracusa, Syracuse
  - Casa di Cura Villa Verde S.r.l, Taranto
  - Ospedale Civile Giuseppe Mazzini, Teramo
  - A.O.U. Città della Salute e della Scienza di Torino, Presidio ospedaliero Molinette, Torino
  - Ospedale Humanitas Gardenigo, Torino
  - Ospedale San Giovanni Bosco ASL Città di Torino, Torino
  - Ospedale San Giovanni Bosco, Torino
  - ASST Bergamo OVEST Ospedale "Treviglio Caravaggio", Treviglio
  - Ospedale di Treviso - ULSS 2 Marca Trevigiana, Treviso
  - Azienda Ospedaliera "Cardinale G. Panico", Tricase
  - Ospedale Maggiore di Trieste, Trieste
  - Santa Maria della Misericordia, Udine
  - Ospedale Castelli di Verbania, Verbania
  - ASP di Vibo Valentia Presidio Ospedaliero "G. Jazzolino", Vibo Valentia
  - Ospedale San Bortolo di Vicenza, Vicenza
  - Ospedale di Oglio Po-ASST di Cremona, Vicomoscano
- Netherlands (27):
  - Ziekenhuis Amstelland, W.L. ten Holt, Amstelven, Amstelveen
  - BovenlJ Ziekenhuis, Cardiology, Amsterdam, Amsterdam
  - Academisch Medisch Centrum, Cardiology, Amsterdam, Amsterdam
  - Rijnstate, Cardiology, Arnhem, Arnhem
  - Rode Kruis Ziekenhuis, Cardiology, Beverwijk, Beverwijk
  - IJsselland Ziekenhuis, Cardiology, Capelle aan den IJssel, Capelle aan den IJssel
  - Van Weel-Bethesda Ziekenhuis, Cardiology, Dirksland, Dirksland
  - Gelderse Vallei Ziekenhuis, Cardiology, Ede, Ede
  - Beatrix Ziekenhuis, Cardiology, Gorinchem, Gorinchem
  - Groene Hart Ziekenhuis, Cardiologie, Gouda, Gouda
  - Zuyderland Medisch Centrum, Cardiologie, Heerlen, Heerlen
  - Elkerliek Ziekenhuis, Cardioloog Bendermacher, P.E.F., Helmond, Helmond
  - Tergooiziekenhuizen, Cardiology, Hilversum, Hilversum
  - Spaarne Gasthuis, Cardiology, Hoofddorp, Hoofddorp
  - Maastricht University Medical Center, Cardiology, Maastricht, Maastricht
  - Isala Diaconessenhuis, Internal Medicine, Meppel, Meppel
  - St. Antonius Ziekenhuis, Cardiology, Nieuwegein, Nieuwegein
  - Radboud Medical Center, Cardiology, Nijmegen, Nijmegen
  - Waterlandziekenhuis, Cardiology, Purmerend, Purmerend
  - Laurentius Ziekenhuis, Cardiology, Roermond, Roermond
  - Franciscus Gasthuis & Vlietland, Cardiology, Rotterdam, Rotterdam
  - Franciscus Gasthuis & Vlietland, Cardiology, Schiedam, Schiedam
  - Franciscus Gasthuis & Vlietland, Neurology, Schiedam, Schiedam
  - HagaZiekenhuis, Sportlaan, Cardio Research, Den Haag, The Hague
  - Cardioloog van de Wal, R.M.A., Uden, Uden
  - Maxima Medisch Centrum, Cardiology, Veldhoven, Veldhoven
  - Streekziekenhuis Koningin Beatrix, Cardiology, Winterswijk, Winterswijk
- Portugal (9):
  - Clínica Vergílio Schneider, Angra do Heroísmo
  - Centro Hospitalar Baixo Vouga, Aveiro
  - Instituto do Coração, Carnaxide
  - Centro Hospitalar Cova da Beira, Covilha
  - Hospital Lusíadas Lisboa, Lisbon
  - Hospital Santa Maria, Lisbon
  - Clínica Cuida Mais, Cuidados de Saúde, Mangualde
  - Centro Hospitalar de Setúbal, Setúbal
  - Centro Hospitalar de Vila Nova de Gaia/Espinho, Vila Nova de Gaia
- Spain (71):
  - Complejo Hospitalrio Universitario A Coruña, A Coruña
  - Hospital General de Albacete, Albacete
  - HM Vallés, Alcalá de Henares
  - Hospital Virgen de Los Lirios, Alcoy
  - Hospital Vega Baja, Alicante
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Del Mar, Barcelona
  - Hospital Universitari de La Vall D´Hebron, Barcelona
  - Hospital Universitario de La Vall D´Hebron, Barcelona
  - Hospital de la San Pau, Barcelona
  - Hospital Madrid Monteprincipe, Boadilla del Monte
  - Hospital Universitario Madrid Montepríncipe, Boadilla del Monte
  - Hospital Universitario de Burgos, Burgos
  - Hospital Carmen Y Severo Ochoa, Cangas del Narcea
  - Hospital General Universitario Santa Lucia, Cartagena
  - Hospital Universitario Santa Lucía, Cartagena
  - Hospital General de Castellón, Castellon
  - Hospital San Pedro de Alcántara, Cáceres
  - Clinica Cardiorreal, Ciudad Real
  - Clínica Cardiologica Dr. Anguita, Córdoba
  - Hospital Virgen de La Luz, Cuenca
  - Hospital Clinico Universitario Virgen de La Arrixaca, El Palmar
  - Hospital Clínico Universitario Virgen de La Arrixaca, El Palmar
  - Hospital Del Vendrell, El Vendrell
  - Hospital General Universitario de Elche, Elche
  - Hospital General Universitario Elda, Elda
  - Hospital de Galdakao-Usansolo, Galdakao
  - Hospital General L'Hospitalet, L'Hospitalet de Llobregat
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat
  - Hospital Perpetuo Socorro, Las Palmas de Gran Canaria
  - Hu de Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria
  - Complejo Asistencial Universitario de León, León
  - Hospital Río Carrión, León
  - Hospital Universitario de La Princesa, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - HM Madrid (H. U. HM Madrid, Cardiology, Madrid 3084), Madrid
  - Hospital San Rafael, Madrid
  - Hu Ramón Y Cajal, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hu La Paz, Madrid
  - Hospital Sanchinaro (H. U. HM Sanchinarro, Cardiology, Madrid 3085), Madrid
  - Hu Puerta de Hierro, Majadahonda
  - Hospital Costa del Sol (Marbella), Marbella
  - Hospital Costa Del Sol, Marbella
  - Hu Virgen de La Victoria, Málaga
  - Hospital Comarcal Medina del Campo, Medina del Campo
  - Hm Puerta Del Sur, Móstoles
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital de La Vega Baja, Orihuela
  - Hospital Son Llàtzer, Palma de Mallorca
  - Clinica Universitaria de Navarra, Pamplona
  - Complejo Hospitlario de Navarra, Pamplona
  - Hospital Virgen Del Camino, Pamplona
  - Hospital El Bierzo, Ponferrada
  - Complexo Hospitalario de Pontevedra, Pontevedra
  - Hospital de Sagunto, Sagunto
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - Hu San Juan de Alicante, Sant Joan de Alacant
  - Hospital Moises Broggi, Sant Joan Despí
  - H. Clinico Univ. de Santiago, Santiago de Compostela
  - Clinica Vida, Seville
  - Consulta Privada, Seville
  - Hospital Virgen Macarena, Seville
  - Hospital Universitario Virgen Del Rocío (Huvr), Seville
  - Hm Torrelodones, Torrelodones
  - Hospital Universitario de Torrevieja, Torrevieja
  - Hospital Clinico Universitario de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Clínico de Valladolid, Valladolid
  - Hospital Universitario de Álava, Vitoria-Gasteiz
- Switzerland (17):
  - Kantonsspital Baden, Innere Medizin, Baden, Baden
  - Praxis Dr. Stefan Kradolfer, Basel, Basel
  - Spital Emmental, Allgemeine Innere Medizin, Burgdorf, Burgdorf
  - Clinique des Grangettes, Dr. Robert Bonvini, Chene-Bougeries, Chêne-Bougeries
  - Université de Fribourg, Département de Médicine,Fribourg, Fribourg
  - Cabinet Dr. Chatelain, Geneve, Geneva
  - Cabinet Dr. Namdar, Geneve, Geneva
  - Praxis PD Dr Sztajzel, Geneva, Geneva
  - Ambulatorio Cardiologia, Dr. Flavio Acquistapace, Lugano, Lugano
  - Cardiocentro Ticino, Cardiologia, Lugano, Lugano
  - Ambulatorio Cardiologia, Dr. Flavio Acquistapace, Manno, Manno
  - Ambulatorio Cardiologia, Dr. Flavio Acquistapace, Mezzovico, Mezzovico
  - Hôpital Neuchâtelois Pourtalès, Neuchâtel, Neuchâtel
  - Praxis Dr. Polikar, Nyon, Nyon
  - Kantonsspital St. Gallen, Sankt Gallen
  - Spitalregion Fuerstenland Toggenburg, Abt. Innere Medizin, Dr. Daniel Nobel, Wil, Wil
  - Universitaetsspital, Rhythmologie, Zuerich, Zurich
- United Kingdom (43):
  - Craigavon Area Hospital, Cardiology, Co. Armagh, Armagh
  - William Harvey Hospital, Geriatric Medicine, Ashford, Ashford
  - Royal Free Hospital, Cardiology, Barnet, Barnet
  - Basingstoke and North Hampshire Hospital, Cardiology, Basingstoke, Basingstoke
  - Ballygomartin Group Practice, Belfast, Belfast
  - The Ulster Hospital, Geriatric Medicine, Belfast, Belfast
  - Belfast City Hospital, Cardiology, Belfast, Belfast
  - Birmingham Heartlands Hospital,Haematology,Birmingham, Birmingham
  - Royal Blackburn Hospital,Cardiology, Blackburn, Blackburn
  - Blackpool Victoria Hospital, Cardiology, Blackpool, Blackpool
  - The Binfield Surgery, Bracknell, Bracknell
  - Westcliffe Medical Practice, Bradford, Bradford
  - Bradford Royal Infirmary, Cardiology, Bradford, Bradford
  - Queen Elizabeth the Queen Mother Hospital, Geriatric Medicine, Margate, Canterbury
  - Carmel Medical Practice, Darlington, Darlington
  - Darent Valley Hospital, Research Office, Cardiology, Dartford, Dartford
  - Russell Hall Hospital,Cardiology, Dudley, Dudley
  - Royal Devon & Exeter Hospital, Geriatric Medicine, Exeter, Exeter
  - Harefield Hospital, Cardiology, Harefield, Harefield
  - Buckinghamshire Healthcare NHS Trust, Cardiology, High Wycombe, High Wycombe
  - Sketty and Killay Medical Centres, Killay, Killay
  - Broadgreen Hospital, Neurology, Liverpool, Liverpool
  - Barts Hospital, Metabolic Medicine, London, London
  - Maryport Health Services, Maryport, Maryport
  - James Cook University Hospital, Cardiology, Middlesbrough, Middlesbrough
  - Royal Gwent Hospital, Dept of Cardiology, Newport, Newport
  - Mowbray House Surgery,Northallerton, Northallerton
  - Danes Camp Medical Practice, Dr. Zafar, Northampton, Northampton
  - Norfolk and Norwich Hospital, Stroke Medicine, Norwich, Norwich
  - Nottingham University Hospitals City Campus, Nottingham, Nottingham
  - Alverton Practice, Penzance, Penzance
  - Peterborough City Hopsital, Cardiology, Peterborough, Peterborough
  - Wansford and Kings Cliffe Practice, Peterborough, Peterborough
  - Pickering Medical Practice, Pickering, Pickering
  - Whiston Hospital, Cardiology, Prescot, Prescot
  - Queen's Hospital, Cardiology, Romford, Romford
  - Lister Hospital, Cardiology, Stevenage, Stevenage
  - Stokesley Health Centre, Stokesley, Stokesley
  - Sunderland Royal Hospital, Cardiology, Sunderland, Sunderland
  - Vine Medical Group, Forest End Site, Waterlooville, Waterlooville
  - Whitby Group Practice, Whitby, Whitby
  - Sleights and Sandsend Medical Practice, Whitby, Whitby
  - Royal Albert Edward Infirmary, Haematology, Wigan, Wigan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Background] Giugliano RP, Ruff CT, Braunwald E, Murphy SA, Wiviott SD, Halperin JL, Waldo AL, Ezekowitz MD, Weitz JI, Spinar J, Ruzyllo W, Ruda M, Koretsune Y, Betcher J, Shi M, Grip LT, Patel SP, Patel I, Hanyok JJ, Mercuri M, Antman EM; ENGAGE AF-TIMI 48 Investigators. Edoxaban versus warfarin in patients with atrial fibrillation. N Engl J Med. 2013 Nov 28;369(22):2093-104. doi: 10.1056/NEJMoa1310907. Epub 2013 Nov 19. PMID 24251359
- [Derived] De Caterina R, Unverdorben M, Chen C, Choi EK, Koretsune Y, Morrone D, Pecen L, Bramlage P, Wang CC, Yamashita T, Kirchhof P. Two-Year Follow-Up of Patients With Atrial Fibrillation Receiving Edoxaban in Routine Clinical Practice: Results From the Global ETNA-AF Program. Clin Cardiol. 2025 Feb;48(3):e70091. doi: 10.1002/clc.70091. PMID 40014354
- [Derived] de Vries TAC, Hemels MEW, Cools F, Crijns HJGM, Yperzeele L, Vanacker P, Blankoff I, Lancellotti P, Mairesse GH, de Veer A, Casado Arroyo R, Catez E, de Pauw M, Vanassche T, de Asmundis C, Kirchhof P, De Caterina R, de Groot JR; ETNA-AF-Europe principal investigators from Belgium and the Netherlands*. Characteristics of patients with atrial fibrillation prescribed edoxaban in Belgium and the Netherlands: insights from the ETNA-AF-Europe study. Neth Heart J. 2021 Mar;29(3):158-167. doi: 10.1007/s12471-020-01518-7. Epub 2021 Jan 7. PMID 33411231
- [Derived] de Vries TAC, Hemels MEW, Cools F, Crijns HJGM, Yperzeele L, Vanacker P, Blankoff I, Lancellotti P, Mairesse GH, de Veer A, Casado Arroyo R, Catez E, de Pauw M, Vanassche T, de Asmundis C, Kirchhof P, De Caterina R, de Groot JR; ETNA-AF-Europe principal investigators from Belgium and the Netherlands. Characteristics of patients with atrial fibrillation prescribed edoxaban in Belgium and The Netherlands: insights from the ETNA-AF-Europe study. Acta Cardiol. 2021 Jun;76(4):431-439. doi: 10.1080/00015385.2020.1746095. Epub 2021 Jan 7. PMID 33406996
- [Derived] De Caterina R, Kelly P, Monteiro P, Deharo JC, de Asmundis C, Lopez-de-Sa E, Weiss TW, Waltenberger J, Steffel J, de Groot JR, Levy P, Bakhai A, Zierhut W, Laeis P, Kerschnitzki M, Reimitz PE, Kirchhof P; ETNA-AF-Europe investigators. Characteristics of patients initiated on edoxaban in Europe: baseline data from edoxaban treatment in routine clinical practice for patients with atrial fibrillation (AF) in Europe (ETNA-AF-Europe). BMC Cardiovasc Disord. 2019 Jul 12;19(1):165. doi: 10.1186/s12872-019-1144-x. PMID 31299906
- [Derived] De Caterina R, Kelly P, Monteiro P, Deharo JC, de Asmundis C, Lopez-de-Sa E, Weiss TW, Waltenberger J, Steffel J, de Groot JR, Levy P, Bakhai A, Zierhut W, Laeis P, Reimitz PE, Kirchhof P; ETNA-AF-Europe investigators. Design and rationale of the Edoxaban Treatment in routiNe clinical prActice for patients with Atrial Fibrillation in Europe (ETNA-AF-Europe) study. J Cardiovasc Med (Hagerstown). 2019 Feb;20(2):97-104. doi: 10.2459/JCM.0000000000000737. PMID 30540648